CLINICAL TRIAL: NCT00543348
Title: A Randomised-Controlled Study Comparing the Peripheral Cutting BalloonTM (Boston Scientific Co.) With a High Pressure Balloon for the Treatment of Arteriovenous Fistula Stenoses
Brief Title: RCT of the Cutting Balloon Versus a High Pressure Balloon for the Treatment of Arteriovenous Fistula Stenoses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, loay kabbani, MD, Vascular Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFHIRB4244
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Stenosis
Keywords: BALLOON ANGIOPLASTY; AUTOGENOUS FISTULA
MeSH Terms: conditions — Constriction, Pathologic | interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): CUTTING BALLOON ANGIOPLASTY
  Interventions: Procedure: CUTTING BALLOON ANGIOPLASTY
- 2 (Placebo Comparator): Balloon angioplasty with a high pressure balloon
  Interventions: Procedure: CUTTING BALLOON ANGIOPLASTY; Procedure: Balloon angioplasty

INTERVENTIONS:
Procedure: CUTTING BALLOON ANGIOPLASTY — CUTTING BALLOON
Procedure: Balloon angioplasty — HIGH PRESSURE BALLOON
  Arms: 2

SUMMARY:
The proposed study will investigate the efficacy of the peripheral cutting balloon (PBC) compared to the high pressure balloon in dilating venous stenosis in hemodialysis fistulas.

2. SPECIFIC AIMS

Study endpoints will be:

Primary Endpoint

1. Primary and assisted patency at 6 months

Secondary Endpoints:

1. Procedure effectiveness/residual stenosis
2. Procedure-related complications
3. Primary patency and primary assisted patency 12 months
4. Secondary patency at 6 and 12 months
5. Number/type of secondary interventions.

ELIGIBILITY:
Inclusion Criteria:

* Dysfunctional fistulas will be recruited based on the presence of clinical and hemodialysis parameters

Exclusion Criteria:

* Arteriovenous prosthetic grafts

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2008-03 (Estimated); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Primary and assisted patency | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GEORGES HADDAD, MD, FACS, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States